CLINICAL TRIAL: NCT04327115
Title: ACTI-PACT : Programme d'ACcompagnement à l'acTIvité Physique Chez la Personne Âgée de 75 Ans et Plus, hospitalisée en CourT séjour gériatrique
Brief Title: Study of an Physical Exercise Program on Older People of 75 Years Old and More, Hospitalized in Geriatric Short Stay
Acronym: ACTI-PACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A01800-57
Record Dates: First submitted 2020-03-23; First posted 2020-03-30 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Physical Activity; Aged
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: stepped wedge cluster randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Other): (C-I-I-I) : the centers apply the "Control" strategy in Period 1 and then apply the "Intervention" strategy in Periods 2 to 4.
  Interventions: Procedure: "Control" strategy; Procedure: "Intervention" strategy
- Arm 2 (Other): (C-C-I-I) : the centers apply the "Control" strategy in periods 1 and 2 and then apply the "Intervention" strategy in periods 3 and 4.
  Interventions: Procedure: "Control" strategy; Procedure: "Intervention" strategy
- Arm 3 (Other): (C-C-C-I) : the centers apply the "Control" strategy in periods 1, 2 and 3 and then apply the "Intervention" strategy for period 4.
  Interventions: Procedure: "Control" strategy; Procedure: "Intervention" strategy

INTERVENTIONS:
Procedure: "Control" strategy — Patients included in the "control" group will received the usual cares of the unit during their stay : support in the gestures of daily life and walking according to their ability and at the discretion of the care teams.
Procedure: "Intervention" strategy — Patients included in the "intervention" group will received the usual cares of the unit during their stay : support in the gestures of daily life and walking according to their ability and at the discretion of the care teams.
  They will also get a physical activity program realized with a nurse or a nursing assistant, twice a day (morning and evening) for 5 days. The intervention consists of physical support with mimed instructions, the nature of which depends on the falling risk of the participant :
  * High falling risk : "out of bed" exercise (on a chair for at least 30 min)
  * Mild falling risk : "out of bed" exercise + "in front of chair" (The participant stands standing in static equilibrium to a chair holding the back of it for 2 minutes, on both feet or one foot)
  * Low falling risk : "out of bed" exercise + "in front of chair" + FTSS exercise (The participant performs a transfer activity of sitting to standing repeated 5 times, with physical assistance or not)

SUMMARY:
The main objective is to assess the effect, compared to usual care, of a nursing accompaniment or nursing assistant intervention in the physical activity of patients hospitalized in the geriatric stay, on the daily number of steps.

The secondary objectives consist in evaluating the effect, compared to usual care, of a nursing or nursing assistant's intervention in physical activity of elderly patients hospitalized on a short geriatric stay in terms of:

* The change of the daily physical exertion in metabolic equivalent
* The change of the daily number of steps
* The change of care course
* The change of in falls occurrence
* The change of autonomy patient
* The change of travels habits

DETAILED DESCRIPTION:
The aging of the French population leads to a significant increase in elderly hospitalizations. These patients are often dependent, polymorbid and precarious from a medical, social and economic point of view, bringing them into a frailty process to which the health system is trying to adapt. In fact, the absence of specific care adapted to frail elderly patients results in an increased risk of functional maladjustment. It is characterized by a loss, during hospitalization, of the ability to perform the activities of daily living alone and a decrease in physical activity. This maladjustment can differ or even prevent return home, increases the risk of falling, the length of stay and health expenses.

The concept of frailty in the elderly is mainly based on the concept of physical vulnerability, and in particular muscular vulnerability. Increasing attention is therefore being paid to physical activity in the elderly, which can prevent the process of maladjustment.

The 2004802 Decree of July 29, 2004 recalls that nurses lift patients and help them to walk without using rehabilitation techniques, to ensure their comfort. The interest of such an approach has already been reported, especially in primary care where nursing support allows a sustained and lasting increase in physical activity in the elderly. To the best of the investigators' knowledge, the effectiveness of such a nursing approach to physical activity support has not been studied in hospitals yet.

The investigators looked for exercises simple, fast and adapted to an elderly population with a very diverse functional maladjustment. The selected intervention is a physical activity based on the activities of daily living to improve postural balance and strengthening the muscles of the lower limbs. This intervention follows the main principles of the latest recommendations of the French High Authority for Health on the elderly fall prevention. It resumes acts such as sitting or standing on a foot corresponding to static equilibrium conditions. It also proposes carrying out transfers from a sitting to standing position and from a standing to sitting position corresponding to motor acts for the lower limbs.

The investigators hypothesize that formalized paramedical support in a geriatric short-stay service prevents the elderly from decreasing their physical activity, and prevents the occurrence of falls and early re-hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 75 years old
* Hospitalization in geriatric short stay
* Informed and express (oral) consent to participate in the study by the patient or the patient's representative
* Affiliation to French Social Security.

Exclusion Criteria:

* Neurological or orthopedic pathology that prevents the performance of one or more exercises corresponding to the patient's level of risk of falling
* Short expected hospital stay
* Contraindication to physical activity
* Person subject to a safeguard of justice measure
* Patient who previously participated to the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in the number of steps | this outcome is assessed at Day 5 after inclusion.
  the relative evolution of the number of steps between the 1st day (D1) and the 5th day (D5) is calculated with this formula : Δ nbsteps (%) = (D5 number of steps - D1 number of steps)*100 / ((D1 number of steps + D5 number of steps)/2).

SECONDARY OUTCOMES:
Change in the daily physical expenditure in metabolic equivalent | This outcome is assessed between Day 1 and Day 5.
  The daily physical expenditure is evaluated by the actimeter in MET (Metabolic Equivalent of Task)
Change in the daily number of steps | This outcome is assessed between Day 1 and Day 5.
  The daily number of steps is evaluated by the actimeter
Change in the daily physical expenditure | This outcome is assessed between Day 1 and Day 5.
  The daily physical expenditure is evaluated by the actimeter
Change in care course | This outcome is assessed between Day 0 and Day 60.
  The care course is evaluated by the length of hospitalization
Change in care course | This outcome is assessed between Day 6 and Day 30.
  The care course is assessed by the occurrence of a new hospitalization
Change in falls occurrence | This outcomes is assessed between Day 0 and Day 6, then while the 60 days after inclusion.
  The falls occurrence is assessed by the number of falls reported by the participant
Change in patient autonomy | This outcomes is assessed at baseline and 60 days after inclusion.
  Autonomy is assessed with Activities of Daily Living (ADL) score. ADL is an autonomy assessment grid (from 0 to 6) for basic activities of daily living (ADL). The lower the score, the more dependent the patient is.
Change in moving habits | This outcomes is assessed at baseline and 60 days after inclusion.
  Moving habits are assessed with the Life-Space Assessment questionnaire. 120 is the highest score (the best mobility) 0 is the worst score (the worst mobility)

CONTACTS AND LOCATIONS:
Locations (1):
- Cédric ANNWEILER , MD, PhD, Angers, France